CLINICAL TRIAL: NCT02477358
Title: The Use of Platelet Rich Fibrin in Pulpal and Periodontal Regeneration in Mature Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0443-14-FB
Record Dates: First submitted 2015-05-26; First posted 2015-06-22 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Pulpal Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: Multiple teeth (2-6 teeth per participant) will be removed with the root attached and then half of the total teeth(per participant) will be placed back in the socket with Platelet Rich Fibrin (PRF) and the other half will be placed in the socket without PRF.
Who Masked: Participant, Care Provider
Masking Description: Participant and Operating Surgeon were masked to tooth designation. Principal investigator/outcomes assessor aware of designation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF Treated (Experimental): Subjects will be randomized to either receive either left tooth platelet rich fibrin; right tooth implant alone, OR right tooth platelet rich fibrin; left tooth implant alone. Following treatment each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
  Interventions: Procedure: Left Tooth Platelet Rich Fibrin; Right Tooth Implant Alone; Procedure: Right Tooth Platelet Rich Fibrin; Left Tooth Implant Alone
- Control (No Intervention): Subjects will be randomized to either receive either left tooth platelet rich fibrin; right tooth implant alone, OR right tooth platelet rich fibrin; left tooth implant alone. Following treatment each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.

INTERVENTIONS:
Procedure: Left Tooth Platelet Rich Fibrin; Right Tooth Implant Alone — All study participants will have two teeth extracted and 2 mm of root removed. Half of the subjects will have platelet rich fibrin endodontic revascularization therapy will be applied to the left tooth socket only. The right tooth is implanted alone. Each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
  Arms: PRF Treated
Procedure: Right Tooth Platelet Rich Fibrin; Left Tooth Implant Alone — All study participants will have two teeth extracted and 2 mm of root removed. Half of the subjects will have platelet rich fibrin endodontic revascularization therapy to the right tooth socket only. The left tooth is implanted alone. Each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
  Arms: PRF Treated

SUMMARY:
In cases of permanent tooth avulsion, it is widely accepted that some necrosis always occurs after avulsion injury. If the pulp tissue does not revascularize or if endodontic therapy is not performed, the pulp space can become infected. Platelet rich fibrin (PRF) is a second generation platelet concentrate that allows the clinician to obtain fibrin membranes enriched with platelets and growth factors from an anticoagulant-free blood harvest. Clinical relevance of PRF and revascularization has been demonstrated in several case studies of avulsion. To date no human clinical trials have been performed evaluating the effectiveness of PRF on pulpal revascularization after reimplantation and its benefits in limiting inflammation. The following study consists of two phases: Phase 1: An in vitro model evaluating the effects of PRF in limiting inflammatory response of pdl cell cultures in the presence of an inflammatory mediators. Phase 2: An in vivo model utilizing mature teeth previously treatment planned for extraction, treating with PRF, reimplanting teeth and following for three to four months before extracting and performing histological analysis. If PRF is capable of promoting revascularization in mature teeth the potential benefits extend to limiting the need for endodontic therapy following mature tooth avulsion, potential for mature tooth transplantation in situations of congenitally missing teeth, and utilization of PRF in endodontic revascularization therapy.

DETAILED DESCRIPTION:
When a tooth is avulsed, it is separated from its socket causing damage to the attachment apparatus. The periodontal ligament (pdl) is a group of specialized connective tissue fibers that attaches the cementum of the root (outer layer) to the alveolar bone. Avulsion can cause damage to the pdl and possible cemental tears. If the periodontal ligament is left attached to the root and minimal time lapse occurs damage to the tissues is usually limited. In these cases, reimplantation is a widely accepted treatment; however the long term success of an avulsed tooth is dependent on various factors. When excessive drying occurs prior to re-implantation, a severe inflammatory response is elicited directly on the root surface which may result in osseous replacement or replacement resorption. Some necrosis always occurs after avulsion injury, and while the necrotic pulp is of little consequence, this necrotic tissue is at high risk for bacterial contamination. If the pulp tissue does not revascularize or if endodontic therapy is not performed, the pulp space can become infected. It has been suggested that treatment strategies should attempt to limit peri-radicular inflammation therefore promoting favorable cemental healing and limiting unfavorable osseous replacement.

Platelet rich fibrin (PRF) is a second generation platelet concentrate that allows the clinician to obtain fibrin membranes enriched with platelets and growth factors from an anticoagulant-free blood harvest and without the addition of artificial biochemical modification. PRF has demonstrated clinical relevance through its ability to stimulate cell proliferation of osteoblasts, gingival fibroblasts, and periodontal ligament (PDL) cells. In addition, PRF has been shown to limit epithelial cell growth therefore promoting connective tissue and alveolar bone regeneration and inhibiting epithelial proliferation. These properties make it a favorable product for surgical procedures requiring micro vascularization.

In vitro studies with PRF and canine dental pulp cells demonstrate PRF's ability to promote chemotaxis and proliferation of the pulp cells and contributed to pulp repair. When PRF was combined with human dental pulp cells derived from extracted third molars it did not interfere with vitality and stimulated proliferation and differentiation. Additionally it upregulated the expression of osteoprotegerin and alkaline phosphatase.

Animal models evaluated PRF granules combined with human pdl stem cells and placed them on the root surface of freshly extracted canine teeth. The teeth were then reimplanted and evaluated histologically after a healing phase. A regeneration of the PDL-like tissue and reduction in ankylosis and inflammation were noted in animals with the PRF granules.

Clinical relevance of PRF and revascularization has been demonstrated in several case studies of avulsion. These case studies utilized a general protocol of minimally instrumenting the avulsed tooth. One study performed a 3 mm resection of the root apex followed by minimal instrumentation of the canal. Blood is then drawn from the patient and PRF is prepared via Choukroun's method. The PRF is then placed on the root surface and condensed into the canal. The tooth was then reimplanted, splinted, and the patient followed for up to 24 months. The tooth tested vital to thermal and percussion testing and radiographically did not show signs of replacement resorption or inflammation.

To date no human studies have been performed evaluating the effectiveness of PRF on pulpal revascularization after reimplantation and its benefits in limiting inflammation. Additionally, only histological evidence of the benefits of PRF has been demonstrated in animal models. If PRF is capable of promoting revascularization in mature teeth the potential benefits extend to limiting the need for endodontic therapy following mature tooth avulsion, potential for mature tooth transplantation in situations of congenitally missing teeth, and utilization of PRF in endodontic revascularization therapy.

The following research would consist of two phases: Phase 1. An in vitro model evaluating the effects of PRF in limiting inflammatory response of pulp and pdl cell cultures in the presence of an inflammatory mediators. Phase 2. An in vivo model utilizing mature teeth previously treatment planned for extraction, treating in accordance to the procedure documented by one group, reimplanting teeth and following for three to four months before extracting and performing histological analysis.

ELIGIBILITY:
Inclusion Criteria:

* any adult with single rooted vital teeth previously treatment planned for extraction to meet their prosthetic or orthodontic needs.

Exclusion Criteria:

* exclusion criteria will include: individuals with systemic illnesses that could compromise vascularity or healing,
* patients who are pregnant,
* or bisphosphonates.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth L Easley, DMD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient's were recruited from the UNMC Dental School
Pre-assignment Details: No pre-assignment details were completed prior to assignment to an arm/group
Units Other Than Participants: Teeth
Groups:
- PRF Treatment; No Treatment: All study participants are scheduled for teeth extraction. Subjects will be randomized to either receive either left tooth PRF; right tooth reimplantation, OR right tooth PRF; left tooth reimplantation. Following treatment each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
  All study participants will have two teeth extracted and 2 mm of root removed. Half of the subjects teeth will have PRF endodontic revascularization therapy and the other teeth will be reimplanted alone. Each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
Period: Overall Study
Arm/Group | PRF Treatment | No Treatment
Started | 18; 36 Teeth | 18; 36 Teeth
Completed (2 teeth (1 Treatment and 1 control) were withdrawn from the study due to early removal and excluded from statistical data.) | 18; 35 Teeth | 18; 35 Teeth
Not Completed | 0; 1 Teeth | 0; 1 Teeth

BASELINE CHARACTERISTICS:
Population: Half of the subjects teeth will have PRF endodontic revascularization therapy and the other teeth will be reimplanted alone.
Units Other Than Participants: Teeth
Groups:
- PRF Treatment: All study participants are scheduled for teeth extraction (between 2 to 6 teeth per participant). Subjects will be randomized to either receive either left tooth PRF; right tooth re-implantation, OR right tooth PRF; left tooth re implantation. Following treatment each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for at least 3 months (up to 11 months) and then tested for vitality before extracting and examining histologically.
  All study participants will have two teeth extracted and 2 mm of root removed. Half of the subjects teeth will have PRF endodontic revascularization therapy. Each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
- No Treatment: All study participants are scheduled for teeth extraction (between 2 to 6 teeth per participant). Subjects will be randomized to either receive either left tooth PRF; right tooth re-implantation, OR right tooth PRF; left tooth re-implantation. Following treatment each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months (up to 11 months) and then tested for vitality before extracting and examining histologically.
  All study participants will have two teeth extracted and 2 mm of root removed. Half of the subjects teeth will be re implanted alone. Each tooth is replaced and splinted to the adjacent teeth. Teeth are followed for 3 months and then tested for vitality before extracting and examining histologically.
- Total: Total of all reporting groups
Arm/Group | PRF Treatment | No Treatment | Total
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (Teeth) | 35 | 35 | 70
Age, Continuous [Median (Full Range); unit: years] — Unit of measure- years
  years | 58.5 [41 to 76] | 58.5 [41 to 76] | 58.5 [41 to 76]
Sex: Female, Male [Count of Units; unit: Teeth] — Population: Units were not evenly split between male/female gender. A larger proportion of total units were measured in male participants.
  Teeth
    Female | 17 | 17 | 34
    Male | 18 | 18 | 36
Pre-treatment Tooth Vitality to Thermal and Percussion Sensitivity [Mean (Standard Deviation); unit: Teeth] — Evaluation recorded to determine the initial vitality of each tooth using Thermal and Percussion Sensitivity
  Teeth
    Pre Thermal | .852 (.089) | .939 (.048) | .8955 (.0685)
    Pre Percussion | .121 (.066) | .092 (.056) | .1065 (.061)
Pre-treatment Tooth Vitality to Electric Pulp Test (EPT) [Mean (Standard Deviation); unit: EPT Units (0-80)] — Evaluation recorded to determine the initial vitality of each tooth using a Electronic Pulp Test (EPT) 0-80 units. There is no specific number that suggests vital vs un-vital but rather it is a trend towards unvital which is determined as 80.
  EPT Units (0-80) | 34.0 (3.0) | 33.1 (3.0) | 33.5 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Vitality of Teeth (Units) Using Thermal and Percussion Sensitivity Trend Observed During Study Duration (3-11 Months)
Description: Teeth (units) measuring vital via the following tests: thermal, percussion. Thermal was utilized with endo cold spray and percussion from tapping on teeth with mouth mirror.
Time Frame: 3-11 months. Each participant was measured for as long as it took to complete their prosthesis. The minimum study duration was 3 months and the maximum duration was 11 months in one subject.
Population: Half of the subjects teeth will have PRF endodontic revascularization therapy and the other teeth will be reimplanted only without PRF endodontic reveascularization therapy.
Measure: Mean (Standard Deviation); unit: Teeth
Units Other Than Participants: Teeth
Groups:
- Experimental: PRF Treated: Teeth Extracted and reimplanted after PRF endodontic revascularization therapy. Splinted to adjacent teeth. Monitored for 3 months then tested for vitality (EPT, Thermal, Percussion), extracted, histologically examined.
- No Intervention: Control: Teeth Extracted and reimplanted. Splinted to adjacent teeth. Monitored for 3 months then tested for vitality (EPT, Thermal, Percussion), extracted, histologically examined.
Arm/Group | Experimental: PRF Treated | No Intervention: Control
Number analyzed (Participants) | 18 | 18
Number analyzed (Teeth) | 35 | 35
Teeth
  Teeth with Thermal Sensitivity Results | .559 (.120) | .592 (.118)
  Teeth with Percussion Sensitivity Results | .065 (.046) | .040 (.034)

2. Primary Outcome: Vitality of Teeth Using Electronic Pulp Test (EPT Units) Trend Observed During Study Duration (3-11 Months)
Description: Teeth (units) measuring vital via the following tests: EPT utilizing EPT units (0-80). There is no specific number that suggests vital vs un-vital but rather it is a trend towards un-vital which is determined as 80.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: EPT Units (0-80)
Units Other Than Participants: Teeth
Arm/Group | PRF Treated | Control
Number analyzed (Participants) | 18 | 18
Number analyzed (Teeth) | 35 | 35
EPT Units (0-80) | 57 (3.79) | 55.45 (3.81)

ADVERSE EVENTS:
Time Frame: Initiation of study to termination of study (11 months total)
Arm/Group | Experimental: PRF Treated | No Intervention: Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
Limitations of study include bias in patient reporting of sensation for vitality testing, lack of control of possible contributing factors including bruxism, and finally differing values for time out of mouth for control vs experimental groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No